CLINICAL TRIAL: NCT01151683
Title: Effects of Magnesium Supplementation on Vascular Structure and Function in Hypertensive Patients
Acronym: MG600
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Mario Fritsch Neves, Full Professor, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MG600
Record Dates: First submitted 2010-06-25; First posted 2010-06-28 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Hypertension; Endothelial Dysfunction
Keywords: hypertension; endothelial dysfunction
MeSH Terms: conditions — Hypertension | interventions — Magnesium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnesium (Active Comparator): Magnesium chelate 600 mg per day
  Interventions: Dietary Supplement: magnesium
- Placebo (Placebo Comparator): Placebo 4 capsules per day
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: magnesium — Magnesium chelate, 300mg (2 capsules of 150mg) twice a day, per oral Total of 600mg per day
  Other Names: Mg supplement
  Arms: Magnesium
Dietary Supplement: placebo — Two capsules of placebo per oral twice a day
  Other Names: Inactive component
  Arms: Placebo

SUMMARY:
Introduction: Magnesium has been the target for many experimental and clinical studies due to the negative correlation between its serum and intracellular levels and the prevalence of hypertension and other cardiovascular diseases.

Objective: To evaluate the effects of magnesium supplementation in hypertensive patients who are under diuretic treatment, including correlation of clinical and nutritional parameters with structural and functional aspects of the macrocirculation.

Methods: A prospective, randomized, double blind, placebo controlled study will be performed in hypertensive patients, aged between 40 and 65 years-old, in regular use of thiazidic diuretic as antihypertensive monotherapy,. The patients will be divided in two main groups according to supplementation with placebo or magnesium chelate 300mg twice a day (total of 600mg magnesium element per day). Before and after 3 and 6 months of supplementation, the patients will be submitted to clinical and nutritional evaluation, biochemical analysis, including intracellular magnesium measurement, and study of the macrocirculation with ambulatory blood pressure monitoring, analysis of flow-mediated dilation of brachial artery, measurement of carotid intima-media thickness, and carotid-femoral and carotid-radial pulse wave velocity to estimate central and peripheral arterial stiffness.

Analysis: Data will be expressed as mean±epm. Statistical analysis will be performed using software Prism® (GraphPad, version 5.0). Continuous variables in each group will be compared using "t test", and P<0.05 will be considered statistically significant.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate whether magnesium supplementation is associated with improved blood pressure control and whether it has beneficial effects on the vascular structure and function in non-diabetic hypertensive patients who are receiving r diuretic therapy.

Patients will be evaluated in a prospective, randomized, double-blind study and will be admitted to the study if they reach all the inclusion criteria and no exclusion criteria.

In this study, magnesium chelate was chosen because of its better absorption rate. The dosages are different in many protocols but in this project the patients will receive 600 mg of magnesium element daily divided in 300 mg twice a day. The patients will be divided in two main groups according to supplementation with placebo or magnesium chelate 300mg twice a day (total of 600mg magnesium element per day). Before and after 3 and 6 months of supplementation, the patients will be submitted to clinical and nutritional evaluation, biochemical analysis, including intracellular magnesium measurement, and study of the macrocirculation with ambulatory blood pressure monitoring, analysis of flow-mediated dilation of brachial artery, measurement of carotid intima-media thickness, and carotid-femoral and carotid-radial pulse wave velocity to estimate central and peripheral arterial stiffness.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 40 and 65 years-old
* Hypertension with mild blood pressure elevation:

  * Systolic BP between 140 and 159mmHg AND/OR
  * Diastolic BP between 90 and 99 mmHg
* Antihypertensive monotherapy with daily use of thiazidic diuretic, at least in the last 30 days
* Signature of the Informed Consent by the patient or his legal representative

Exclusion Criteria:

* Evidences for secondary hypertension
* Hypertension in stage 2, SBP ≥ 160mmHg and/or DBP ≥ 100mmHg, before the beginning of supplementation
* Blood pressure > 180 x 100 mmHg in any phase of the study
* Body mass index > 35 kg/m2
* Diabetes Mellitus
* Renal disease presenting glomerular filtration rate < 60ml/min
* Coronary artery disease clinically evident with previous episode of myocardial infarction and/or myocardial revascularization
* Clinical signs of heart failure
* History of stroke
* Any condition, disease or therapy that, under investigator's opinion, may influence objectives, results, or put in risk the safety of the patients.
* Pregnancy
* Patients should not be taking any mineral or vitamin supplements
* Gastrointestinal conditions

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Improvement of vascular function | six months

SECONDARY OUTCOMES:
Improvement of vascular structure and blood pressure | six months

CONTACTS AND LOCATIONS:
Overall Officials: Mario F Neves, MD, PhD, Principal Investigator — State University of Rio de Janeiro
Locations (1):
- Department of Clinical Medicine, State University of Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Cunha AR, Medeiros F, Umbelino B, Oigman W, Touyz RM, Neves MF. Altered vascular structure and wave reflection in hypertensive women with low magnesium levels. J Am Soc Hypertens. 2013 Sep-Oct;7(5):344-52. doi: 10.1016/j.jash.2013.04.008. Epub 2013 Jun 2. PMID 23735418